CLINICAL TRIAL: NCT06066710
Title: Trial of Propranolol in Older Adults with Primary Progressive Aphasia
Brief Title: Propranolol in Primary Progressive Aphasia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, David Beversdorf, Professor, Department of Radiology & Thompson Center for Autism & Neurodevelopmental Disorders, University of Missouri-Columbia, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2097152
Record Dates: First submitted 2023-09-08; First posted 2023-10-04 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Aphasia, Primary Progressive
MeSH Terms: conditions — Aphasia, Primary Progressive | interventions — Propranolol; Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propanolol and MRI (Experimental): Participants will receive propranolol via oral capsule. The drug dosage will be titrated slowly to ensure the drug is tolerated well.
  Interventions: Drug: Propranolol; Device: Magnetic Resonance Imaging (MRI)
- Placebo and MRI (Placebo Comparator): Participants will receive placebo via oral capsule.
  Interventions: Device: Magnetic Resonance Imaging (MRI); Drug: Placebo

INTERVENTIONS:
Drug: Propranolol — Propranolol will be given on a titration schedule in which participants will begin with small doses of the drug and increase to a larger dosage over the course of three weeks. Propranolol will be taken for a total of 9 weeks.
  Arms: Propanolol and MRI
Device: Magnetic Resonance Imaging (MRI) — Magnetic Resonance Imaging (MRI) will be performed at 3 Tesla and 7 Tesla, for both propranolol and placebo arms.
Drug: Placebo — Placebo will be given on the same schedule as the propranolol regime.
  Arms: Placebo and MRI

SUMMARY:
The purpose of this study is to find out how the language of people with Primary Progressive Aphasia is affected by Propranolol. Propranolol is not FDA approved for the treatment of Primary Progressive Aphasia. Propranolol is FDA approved for the treatment of heart conditions such as blood pressure.

This research is being done because there are currently no drug treatment options for language impairments and anxiety often experienced by people with Primary Progressive Aphasia.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 50 and older
* 2. Primary Progressive Aphasia diagnosis
* 3. Native English speaker

Exclusion Criteria:

* 1. Unable to provide consent
* 2. Taking alpha 2 agonists (clonidine and guanfacine)
* 3. Other major psychological or neurological diagnosis
* 4. Major head trauma that contributed to their condition
* 5. Allergic reaction to adhesives
* 6. Uncorrected vision/hearing impairments
* 7. Diabetes
* 8. Reactive airway disease
* 9. Untreated hypothyroidism
* 10. Bradyarrhythmia
* 11. Unexplained syncope
* 12. Pregnancy (assessed verbally on the days of MR imaging)
* 13. Drugs that interact with propranolol, such as alpha 2 agonists
* 14. Claustrophobia, inner ear implants, aneurysm or other surgical clips, metal foreign bodies in eye, pacemaker or other contraindication to MR scanning. Subjects with any implanted device that cannot be verified as MRI compliant will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Neuropsychological Assessment Battery Naming Test | Day 1, 4 Weeks, 8 Weeks, 10 Weeks, 14 Weeks,18 Weeks

SECONDARY OUTCOMES:
Change in State-Trait Anxiety Inventory for Adults | Day 1, 4 Weeks, 8 Weeks, 10 Weeks,14 Weeks,18 Weeks
  The State-Trait Anxiety scores range from 20-40. A higher score indicates more anxiety.
Change in Semantic Word Fluency Tasks | Day 1, 8 Weeks,18 Weeks
  The Semantic Word Fluency task measures the subject's ability to name as many items in a minute in a given category. The total number of correct and non-repeated responses are totaled for each category. There is no minimum or maximum score. Higher scores indicate better word fluency.

CONTACTS AND LOCATIONS:
Overall Officials: David Beversdorf, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mesulam MM. Primary progressive aphasia. Ann Neurol. 2001 Apr;49(4):425-32. PMID 11310619
- [Background] Mesulam M, Weintraub S. Primary progressive aphasia and kindred disorders. Handb Clin Neurol. 2008;89:573-87. doi: 10.1016/S0072-9752(07)01254-7. No abstract available. PMID 18631780
- [Background] Gorno-Tempini ML, Hillis AE, Weintraub S, Kertesz A, Mendez M, Cappa SF, Ogar JM, Rohrer JD, Black S, Boeve BF, Manes F, Dronkers NF, Vandenberghe R, Rascovsky K, Patterson K, Miller BL, Knopman DS, Hodges JR, Mesulam MM, Grossman M. Classification of primary progressive aphasia and its variants. Neurology. 2011 Mar 15;76(11):1006-14. doi: 10.1212/WNL.0b013e31821103e6. Epub 2011 Feb 16. PMID 21325651
- [Background] Johnson JK, Diehl J, Mendez MF, Neuhaus J, Shapira JS, Forman M, Chute DJ, Roberson ED, Pace-Savitsky C, Neumann M, Chow TW, Rosen HJ, Forstl H, Kurz A, Miller BL. Frontotemporal lobar degeneration: demographic characteristics of 353 patients. Arch Neurol. 2005 Jun;62(6):925-30. doi: 10.1001/archneur.62.6.925. PMID 15956163
- [Background] Grossman M. Primary progressive aphasia: clinicopathological correlations. Nat Rev Neurol. 2010 Feb;6(2):88-97. doi: 10.1038/nrneurol.2009.216. PMID 20139998
- [Background] Albert ML, Bachman DL, Morgan A, Helm-Estabrooks N. Pharmacotherapy for aphasia. Neurology. 1988 Jun;38(6):877-9. doi: 10.1212/wnl.38.6.877. PMID 3368068
- [Background] Walker-Batson D, Curtis S, Natarajan R, Ford J, Dronkers N, Salmeron E, Lai J, Unwin DH. A double-blind, placebo-controlled study of the use of amphetamine in the treatment of aphasia. Stroke. 2001 Sep;32(9):2093-8. doi: 10.1161/hs0901.095720. PMID 11546902
- [Background] Beversdorf DQ. Pharmacotherapy of aphasia. J Head Trauma Rehabil. 2007 Jan-Feb;22(1):65-6. doi: 10.1097/00001199-200701000-00008. No abstract available. PMID 17235233
- [Background] Zamzow RM, Ferguson BJ, Stichter JP, Porges EC, Ragsdale AS, Lewis ML, Beversdorf DQ. Effects of propranolol on conversational reciprocity in autism spectrum disorder: a pilot, double-blind, single-dose psychopharmacological challenge study. Psychopharmacology (Berl). 2016 Apr;233(7):1171-8. doi: 10.1007/s00213-015-4199-0. Epub 2016 Jan 14. PMID 26762378
- [Background] Beversdorf DQ, Sharma UK, Phillips NN, Notestine MA, Slivka AP, Friedman NM, Schneider SL, Nagaraja HN, Hillier A. Effect of propranolol on naming in chronic Broca's aphasia with anomia. Neurocase. 2007 Aug;13(4):256-9. doi: 10.1080/13554790701595471. PMID 17886000
- [Background] Faigel HC. The effect of beta blockade on stress-induced cognitive dysfunction in adolescents. Clin Pediatr (Phila). 1991 Jul;30(7):441-5. doi: 10.1177/000992289103000706. PMID 1879101
- [Background] Laverdure B, Boulenger JP. [Beta-blocking drugs and anxiety. A proven therapeutic value]. Encephale. 1991 Sep-Oct;17(5):481-92. French. PMID 1686251
- [Background] Cahana-Amitay D, Albert ML, Pyun SB, Westwood A, Jenkins T, Wolford S, Finley M. Language as a Stressor in Aphasia. Aphasiology. 2011;25(2):593-614. doi: 10.1080/02687038.2010.541469. Epub 2011 Apr 19. PMID 22701271